CLINICAL TRIAL: NCT00611637
Title: A Pilot Clinical Trial of CMV pp65 Specific T Cell Adoptive Immunotherapy in Patients Who Have Undergone Allogeneic Stem Cell Transplantation for Malignant Disease
Brief Title: CMV pp65 Specific T Cell Adoptive Immunotherapy in Allogeneic Stem Cell Transplantation for Malignant Disease
Acronym: CMV-BMT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: H. Kim Lyerly (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, H. Kim Lyerly, Professor, Gen & Thor Surgery, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 4138-07-10R5; IND 11649
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Allogeneic Stem Cell Transplantation
Keywords: Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: CMV pp65 Specific T Cells

INTERVENTIONS:
Biological: CMV pp65 Specific T Cells — Donor derived CMV pp65 specific T cells (1 x 105 CD3+ cells/kg (maximum 1 x 107 CD3+ cells) will be infused into recipient over 10 minutes.

SUMMARY:
The purpose of this study is to determine the safety and feasibility of CMV specific, T cell adoptive immunotherapy in patients who have undergone allogeneic stem cell transplantation for malignant disease.

DETAILED DESCRIPTION:
The primary purpose of this clinical trial is to evaluate the safety of this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Stratum 1: Subjects must be undergoing a non-myeloablative stem cell transplant from a 6/6 matched, sibling donor for the treatment of a malignancy
* Stratum 2: Subjects must be undergoing a non-myeloablative stem cell transplant from a 3/6, 4/6, or 5/6 matched, sibling donor for the treatment of a malignancy.
* Stratum 3: Subjects must be undergoing a myeloablative stem cell transplant from a 3/6, 4/6, or 5/6 matched, sibling donor for the treatment of a malignancy.
* Donor must be CMV sero-positive.
* Karnofsky performance status ≥ 70%.
* Subject and donor must be one of the following HLA types: HLA A*0201, HLA-A*0101, HLA-A*2402, HLA-B*0702, HLA-B*0801, HLA-B*35, HLA-DR*1, or HLA-DR*4.
* Availability of the stem cell donor to provide multiple PBMC samples for T-cell culture if needed. These samples could be obtained via a 90cc peripheral blood draw or through leukapheresis. Stem cell donor must satisfy BMT Program criteria for undergoing leukapheresis to provide DLI and consent to provide repeat leukapheresis if this is necessary.
* Ability to understand and provide signed informed consent that fulfills Institutional Review Board guidelines.
* Ability to return to Duke University Medical Center for adequate follow-up as required by this protocol.
* In order to receive their T cell infusions, subjects should be:
* At least 2 weeks from the time of their allogeneic stem cell transplant.
* Without Grade 3 or 4, non-hematologic, major organ toxicity within the preceding 1 week; all non major organ toxicities must have resolved to grade-2 or less.

Exclusion Criteria:

* Pregnant women and nursing mothers.
* Current or prior history of brain metastases.
* More than 12 months since their allogeneic stem cell re-infusion.
* HIV+, Hepatitis BsAg+, Hepatitis C Ab+

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2005-08; Primary Completion 2008-02 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Number of CMV pp65 specific CD8+ T cells produced. | Pre-infusion.
Development of grade III-IV GVHD or major organ toxicity. | Continuously for 100 days post-transplant.

SECONDARY OUTCOMES:
Presence of CMV in peripheral blood. | Tested before and following transplant and infusion.
Percentage of CD8+ T cells that are CMV pp65 specific. | Assessed weekly up to 6 months following T cell infusion.

CONTACTS AND LOCATIONS:
Overall Officials: H. Kim Lyerly, M.D., Principal Investigator — Duke University; Michael A Morse, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States